CLINICAL TRIAL: NCT03890380
Title: Safety and Performance Evaluation of the Magneto Wire
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Magneto Thrombectomy Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-01
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magneto Wire (Experimental): Patients treated with Magneto Wire
  Interventions: Device: Magneto Wire

INTERVENTIONS:
Device: Magneto Wire — Patients will be treated with Magneto Wire

SUMMARY:
A prospective, open label single arm feasibility study to evaluate the safety and performance of the Magneto Wire in patients diagnosed with acute ischemic stroke and planned for thrombectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within defined timelines.
* Age 18-85 years old
* NIHSS ≥ 8
* No significant pre-stroke functional disability (mRS ≤ 1)

Exclusion Criteria:

* Life expectancy of less than 90 days
* Neurological signs that are rapidly improving prior to or at time of treatment
* NIHSS≥30 or state of coma
* Ongoing seizure
* Current use of cocaine or other vasoactive substance
* Known bleeding diathesis
* Known hemorrhagic or coagulation deficiency
* Evidence of active systemic infection
* Current use of oral anticoagulants INR > 3
* Administration of heparin or Novel Oral Anticoagulants within 48 hours preceding the onset of stroke and have an abnormal aPTT at presentation
* Platelet count < 50,000/mm3
* Glucose <50 mg/dL (2.8 mmol, 2.6mM)
* Uncontrolled hypertension (SBP>185 or DBP>110) refractory to pharmacological management
* Known hypersensitivity or allergy to radiographic contrast agents
* Pregnancy or lactating female
* Subject already enrolled in a clinical study involving experimental medication or device
* CT scan or MRI with evidence of acute intracranial hemorrhage, ASPECT score<6, mass effect and/or intracranial tumor.
* Angiographic evidence of carotid dissection, or high grade stenosis that will prevent access to the clot, or cerebral vasculitis, or intracranial stenosis
* Blood vessel with extreme tortuosity or other conditions preventing the access of the device.
* Angiographic evidence of carotid dissection, complete cervical carotid occlusions or vasculitis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | 24 (±8) hours post procedure
  Occurrence of Device-related Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Safety Assessment | 90 (±10) days
  Occurrence of Device-related Serious Adverse Events (SAEs)
Revascularization | immediate
  Revascularization in the immediate post procedure angiogram, using modified Thrombolysis in Cerebrovascular Infarction (mTIC≥2b)
Distal Embolism | immediate
  Evidence of Infarction of a previously uninvolved vascular territory in the immediate post procedure angiogram
National Institutes of Health Stroke Scale (NIHSS) | 24 (±8) hours post procedure
  NIHSS scale is used to evaluate the severity of a stroke by assessing the stroke-related neurologic deficit. Scores range from 0-42, a higher score indicates a higher severity.
Modified Rankin Scale | 90 (±10) days
  Modified Rankin scale is used to evaluate the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scores range from 0-6 (0-no symptoms, 6- death)

CONTACTS AND LOCATIONS:
Overall Officials: Shally Sharon, Study Director — Magneto Thrombectomy Solutions
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No